CLINICAL TRIAL: NCT04472715
Title: EVALUATION OF THE EFFICACY OF FOLLICULAR UNIT EXTRACTION VERSUS FOLLICULAR UNIT EXTRACTION WITH PLATELETS RICH PLASMA IN TREATMENT OF CICATRICAL ALOPECIA
Brief Title: Hair Transplantation in Cicatricial Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, marwa eldeeb, Lecturer of dermatology, Alexandria University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 00007555
Record Dates: First submitted 2020-07-12; First posted 2020-07-15 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hair Transplantation; Cicatricial Alopecia
Keywords: hair loss, follicuular unit extraction, platelet rich plasma
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- follicular unit extraction (Experimental): extraction of hair follicle unit from donar area and tranplant it into recepient bald area
  Interventions: Procedure: follicular unit extarcation and platelet rich plasma
- foolicular unit extraction and platelet rich plasma (Experimental): the same procedure mentioned above coupled with session of platelet rich plasma before and after transplantation
  Interventions: Procedure: follicular unit extarcation and platelet rich plasma

INTERVENTIONS:
Procedure: follicular unit extarcation and platelet rich plasma — hair transplantation procedure

SUMMARY:
follicular unit extraction as a method of hair transplantation in cicatricial alopecia

DETAILED DESCRIPTION:
The study will include 20 patients with cicatrical alopecia.Patients will be randomly assigned into two groups:Group (A):include ten patients will undergo (FUE) alone.

Group (B): include ten patients will undergo(FUE) and (PRP).3-Surgical technique:

* Preoperative Investigations including complete blood count, coagulation profile and hepatitis viral markers.

  1-Group(A): will undergo (FUE)
* Washing the scalp with antiseptic shampoo before the procedure.
* Tumuscentanaesthesia:The donor area is anesthetized with a lidocaine 1% solution diluted with 20 cc saline in addition to adrenaline.
* Creation of micropunches(0.7-1 mm) using micromotor.
* After removal of the punch,the follicular unit is extracted with Jweler's forceps.
* Extracted grafts are then placed on chilled saline gauze for maximum four hours until ready for transplantation.
* The recipient area is prepared with rectangular scalpel blades 1mm or hypodermic blades 0.9 mm.
* Implantation using fine tipped jweler's forceps.
* Finally, receptor and donor areas will be softly cleansed with saline and crepe bandage is applied.

  2-Group (B): FUE+PRP
* The same procedure will be done but grafts will be placed in Prp solution.
* Prp session one week before transplantation then monthly for 3 monthes after (FUE).
* Preparation of PRP
* 10 cc blood will be aspirated in test tube contained a modified solution of anticoagulant,called acid-citrate-dextrose type (ACDA), in which the physiological pH will reached to preserve the platelet integrity.
* The first spin of whole blood sample will be at 2500 rpm for 4 minutes
* The second spin at 4000 for 20 minutes for obtained plasma.
* Platelets are separated as a pellet at the bottom of the tube from platelet-poor plasma (PPP) above. The platelet-rich pellet is resuspended in remaining amount of plasma. The resulting suspension is used as PRP.
* Prp is injected in the recipient area. 4-Follow up:
* Follow up clinically by digital photographs and trichoscopy 1 week after operation, after 3 months and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with unacceptable visible scarring alopecia.

  * Adequate donor area.
  * patient free of signs of disease activity evidenced by trichoscopy.
  * Patients having inadequate laxity for a strip excision (too tight skin).
  * When previous scars of strip surgeries make further strips impossible.

Exclusion Criteria:

* • Inadequate donor area.

  * Signs of active disease or infection.
  * Patient who is not willing for long sessions for several hours or multiple sessions as needed due to the slowness of the process
  * Contraindications for surgical procedure as bleeding tendency.
  * Contraindications for PRP as (cardiovascular, autoimmune disorders, hematological disorders and neoplasms).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
hair regrowth | 6 months
  transplanted hair develop int new hair growth in bald area

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt